CLINICAL TRIAL: NCT06044831
Title: Evaluating BSW HWC's Population Health Model Expansion at Bonton Farms: A Place-Based Quasi-Experimental Study Linking Medical and Social Services
Brief Title: Expanded Population Health Model Evaluation
Status: Recruiting | Type: Observational
Sponsor: Baylor Research Institute (Other)
Collaborators: Southern Star Medical Research Institute (Unknown)
Responsible Party: Principal Investigator, Kevin Sykes, Director of Clinical Research, Baylor Research Institute
Other Study IDs: Baylor IRB 023-136
Record Dates: First submitted 2023-08-31; First posted 2023-09-21 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Chronic Disease; Quality of Life
Keywords: Life Essential 8; Cardiovascular Disease
MeSH Terms: conditions — Chronic Disease; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Expanded Population Health Access: Participants living in the neighborhood with access to expanded population health model.
  Interventions: Behavioral: Expanded Population Health Model

INTERVENTIONS:
Behavioral: Expanded Population Health Model — This intervention includes the current population health model in addition to expanded programming from a local community organization. The current population health model with Baylor Scott & White Health and Wellness Center includes access to primary care, general wellness programs such as cooking classes and nutritional counseling, and evidence-based disease management and prevention. The additional programs from a local community organization focus on human essentials integral to improving health and quality of life and include: health and wellness, economic stability, safe and affordable housing, transportation, a sense of belonging, education, and access to fair credit.

SUMMARY:
This study will evaluate the impact of a comprehensive wellness and social determinants of health intervention on cardiovascular health in a community setting of the Bonton neighborhood. Participants will not be assigned to intervention activities, but health and wellbeing indicators will be collected in relation to how they choose to participate in activities over the year.

DETAILED DESCRIPTION:
The specific aims of this study are to 1) evaluate whether a population health model integrated into a community setting improves cardiovascular health and quality of life in adults 18 years or older and 2) evaluate which programs and services provide the most impact for specific sub-groups of individuals, e.g., elderly, individuals with diabetes, etc.

Participants will receive programs from the existing population health model from Baylor Scott & White Health and Wellness Center with additional programs from a local community organization. Individuals will complete study measures at baseline, 6 months, and 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Ability to alter diet and/or physical activity
* Willing to participate in a 12-month study
* Willing and able to participate in programs at Bonton Farms
* Cannot have participated in an intensive lifestyle change program (Group Lifestyle Balance, Health Eating and Lifestyle Program, or first cohort of apprenticeship) in the last 6 months or have attended more than two weeks of an intensive lifestyle change program
* Cannot be diagnosed with a terminal illness
* Cannot be pregnant or planning to get pregnant in the next 12 months

Exclusion Criteria:

* Below the age of 18 years
* Unable to alter diet and physical activity due to medical condition
* Not willing to participate in a 12-month study
* Not willing and unable to participate in programs at Bonton Farms
* Participated in an intensive lifestyle change program (Group Lifestyle Balance, Health Eating and Lifestyle Program, or first cohort of Bonton Farms' apprenticeship) or has attended more than two weeks of an intensive lifestyle change
* Be diagnosed with a terminal illness
* Currently pregnant or planning to get pregnant in the next 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Participants living in the neighborhood with access to expanded population health model.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-08-28 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Cardiovascular Health Score | Baseline and 6 Months
  Life's Essential 8 composite score includes 8 metrics used to measure cardiovascular health. The metrics are diet, physical activity, nicotine exposure, sleep health, body mass index, blood lipids, blood glucose, and blood pressure. Each individual metric is scored 0-100 based on clinical thresholds and the composite score is the unweighted, aggregate of all the metrics. Scores 0-49 are considered low cardiovascular health, 50-79 moderate cardiovascular health, and 80-100 high cardiovascular health.
Centers for Disease Control and Prevention Health Related Quality of Life Scale | Baseline and 6 Months
  Measured by self report with Centers for Disease Control and Prevention Health Related Quality of Life Scale. Two modules (Healthy Days and Healthy Days Symptoms) are assessed in 9 items. Only the items in the Healthy Days Module produces a score and it is the sum of healthy and unhealthy days. A higher sum is associated with mental distress or activity limitation.

SECONDARY OUTCOMES:
Cardiovascular Health Score | 12 Months
  Life's Essential 8 composite score includes 8 metrics used to measure cardiovascular health. The metrics are diet, physical activity, nicotine exposure, sleep health, body mass index, blood lipids, blood glucose, and blood pressure. Each individual metric is scored 0-100 based on clinical thresholds and the composite score is the unweighted, aggregate of all the metrics. Scores 0-49 are considered low cardiovascular health, 50-79 moderate cardiovascular health, and 80-100 high cardiovascular health.
Metabolic Syndrome | Baseline, 6 Months, and 12 Months
  Measured by the presence of three or more elevated factors from waist circumference, triglycerides, high density lipoprotein cholesterol, blood pressure, and A1C.
Centers for Disease Control and Prevention Health Related Quality of Life Scale | 12 Months
  Measured by self report with Centers for Disease Control and Prevention Health Related Quality of Life Scale. Two modules (Healthy Days and Healthy Days Symptoms) are assessed in 9 items. Only the items in the Healthy Days Module produces a score and it is the sum of healthy and unhealthy days. A higher sum is associated with mental distress or activity limitation.
Services utilization | Baseline, 6 Months, and 12 Months
  Measured by self-report survey.
Perceived Stress Scale | Baseline, 6 Months, and 12 Months
  Measured by self-report with Perceived Stress Scale with 10 items. Each item is scored 0-4. A higher sum score indicates higher perceived stress.
Center for Epidemiologic Studies Depression Scale 10 | Baseline, 6 Months, and 12 Months
  Measured by self-report with Center for Epidemiologic Studies Depression Scale 10 with 10 items. Each item is scored 0-4. A sum of 10 or higher indicates depressive symptoms.
Medical Outcomes Study Social Support Survey | Baseline, 6 Months, and 12 Months
  Measured by self-report with Medical Outcomes Study Social Support Survey. This instrument includes 4 subscales (Emotional/informational Support, Tangible Support, Affectionate Support, Positive Social Interaction) with 18 items. Each item is scored 1-5. A higher subscale average indicates greater social support. Additionally, an overall support index can also be calculated by taking the average of the 18 items included in subscales and the score for Question 13. A higher score on the overall support index indicates greater social support.
Motivation and Attitudes Toward Changing Health | Baseline, 6 Months, and 12 Months
  Measured by self-report with Motivation and Attitudes Toward Changing Health. This instrument includes 3 subscales (Willingness, Worthwhile, and Ability) with a total of 9 items. Each item is scored 1-5. A higher subscale average indicates one or more of the following: 1) greater willingness to do things to manage health, 2) more likely to view benefits of change as worthwhile, and/or 3) feeling more capable of making and sustaining change.
Brief Resilience Scale | Baseline, 6 Months, and 12 Months
  Measured by self-report with Brief Resilience Scale with 6 items. Each item is scored 1-5. A higher sum score indicate higher resiliency.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin Sykes, PhD, MPH, Principal Investigator — Baylor Scott & White Health and Wellness Center
Locations (1):
- Baylor Scott & White Health and Wellness Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided